CLINICAL TRIAL: NCT04232085
Title: Regenerative Medicine to Restore Hematopoiesis and Immune Function in Immunodeficiencies and Inherited Bone Marrow Failures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Maryland Stem Cell Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B19126; IRB00227401 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2019-12-30; First posted 2020-01-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Primary Immune Deficiency Disorder; Immune Deficiency Disease; Bone Marrow Failure; Short Telomere Length; Fanconi Anemia; Non Fanconi DNA-DSB Repair Disorder; Hoyeraal-Hreidarsson Syndrome; Dyskeratosis Congenita; Telomere Biology Disorder; Short Telomere Syndrome
Keywords: Bone Marrow Transplantation
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Immune Deficiency Disease; Bone Marrow Failure Disorders; Fanconi Anemia; Hoyeraal Hreidarsson syndrome; Dyskeratosis Congenita | interventions — Alemtuzumab; fludarabine; Melphalan; Whole-Body Irradiation; Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: This is a Phase II prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PID/IDS/IBMFS (Experimental): Alemtuzumab IV infusion over 2 hours on days -14, -13, and -12. Day -14 3 mg followed by 10 mg. Day -13 15 mg (or 10 mg if <10 kg). Day -12 20 mg (or 10 mg if <10 kg).
  Fludarabine 30 mg/m2/day IV infusion over 2 hours on days -6 to -2. Melphalan 70 mg/m2/day IV infusion over 30-60 minutes on days -3 and -2. (Or may be given as a single infusion of 140 mg/m2/day on day -2.) Total body irradiation (PID/IDS): 200 cGy will be administered in a single fraction on day -1.
  Bone Marrow will be harvested and infused on day 0. Post-transplantation Cyclophosphamide 50mg/kg will be given on D+3 post-transplant (within 60-72 hr of marrow infusion) and on D+4 post-transplant.
  Tacrolimus begins on day 5, at least 24 hours after completion of posttransplantation Cy at 0.015mg/kg IBW/dose IV over 4 hours every 12 hours.
  Mycophenolic acid mofetil (MMF) begins on day 5 at a dose of 15 mg/kg PO TID (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1 g PO TID).
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Melphalan; Radiation: Low Dose Total Body Irradiation; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Short Telomere Syndrome (Experimental): Alemtuzumab IV infusion over 2 hours on days -14, -13, and -12. Day -14 3 mg followed by 10 mg. Day -13 15 mg (or 10 mg if <10 kg). Day -12 20 mg (or 10 mg if <10 kg).
  Fludarabine 30 mg/m2/day IV infusion over 2 hours on days -6 to -2. TBI 200 cGY day -1 Bone Marrow will be harvested and infused on day 0. Post-transplantation Cyclophosphamide 25-50mg/kg will be given on D+3 post-transplant (within 60-72 hr of marrow infusion) and on D+4 post-transplant. Starting dose for haplo/MMUD= 50 mg/kg; starting dose for HLA matched= 25 mg/kg Tacrolimus begins on day 5, at least 24 hours after completion of post transplantation Cy at 0.015mg/kg IBW/dose IV over 4 hours every 12 hours.
  Mycophenolic acid mofetil (MMF) begins on day 5 at a dose of 15 mg/kg PO TID (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1 g PO TID).
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Radiation: Low Dose Total Body Irradiation; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Fanconi Anemia or DNA-dsb repair (Experimental): Alemtuzumab IV infusion over 2 hours on days -14, -13, and -12. Day -14 3 mg followed by 10 mg. Day -13 15 mg (or 10 mg if <10 kg). Day -12 20 mg (or 10 mg if <10 kg).
  Fludarabine 30 mg/m2/day IV infusion over 2 hours on days -6 to -2. TBI 200 cGY day -1 Bone Marrow will be harvested and infused on day 0. Post-transplantation Cyclophosphamide 25 mg/kg will be given on D+3 post-transplant (within 60-72 hr of marrow infusion) and on D+4 post-transplant.
  Tacrolimus begins on day 5, at least 24 hours after completion of post transplantation Cy at 0.015mg/kg IBW/dose IV over 4 hours every 12 hours.
  Mycophenolic acid mofetil (MMF) begins on day 5 at a dose of 15 mg/kg PO TID (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1 g PO TID).
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Radiation: Low Dose Total Body Irradiation; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Alemtuzumab — Preparative regimen
  Other Names: Campath
Drug: Fludarabine — Preparative regimen
Drug: Melphalan — Preparative regimen
  Arms: PID/IDS/IBMFS
Radiation: Low Dose Total Body Irradiation — Preparative regimen
Drug: Cyclophosphamide — GVHD prophylaxis
  Other Names: Cytoxan
Drug: Tacrolimus — GVHD prophylaxis
  Other Names: FK506, Prograf
Drug: Mycophenolate Mofetil — GVHD prophylaxis
  Other Names: MMF, Cellcept

SUMMARY:
Phase II prospective trial to assess the rates of donor engraftment using reduced intensity conditioning (RIC) hematopoietic stem cell transplant (HSCT) and post-transplant cyclophosphamide (PTCy) for patients with primary immune deficiencies (PID), immune dysregulatory syndromes (IDS), inherited bone marrow failure syndromes (IBMFS), short telomere syndromes, Fanconi anemia, and non-Fanconi DNA double-strand break (DNA-dsb) repair disorder.

DETAILED DESCRIPTION:
Allogeneic blood and marrow transplantation (alloBMT) is the only curative therapy for many primary immune deficiencies (PID), immune dysregulatory syndromes (IDS), and inherited bone marrow failure syndromes (IBMFS). The best reported outcomes are with human leukocyte antigen (HLA)- matched sibling donors, however, only 30% of children in need of a BMT have an HLA-matched sibling. Use of alternative donors has been limited by unacceptably high rates of transplant-related mortality (TRM), graft rejection, infection, and graft-versus-host disease (GVHD). Reduced intensity conditioning (RIC) regimens have been used for this patient population with improved survival and decreased TRM, but graft failure and sustained donor chimerism have emerged as significant obstacles. Thus, there is an urgent need to develop a RIC platform that improves survival and decreases TRM while maximizing donor engraftment, which is essential for cure.

A large and growing body of literature demonstrates that post-transplant cyclophosphamide (PTCy) allows for the safe and effective use of HLA-matched and mismatched related and unrelated donors and haploidentical related donors after RIC alloBMT. PTCy offers a unique opportunity to 1) broaden donor availability, 2) promote durable engraftment of donor cells, 3) achieve low rates of GVHD and TRM, 4) foster robust immune reconstitution and immunity, and 5) shorten the duration of additional post-transplant immune suppression (IS) required to prevent GVHD. The investigators proposed platform is uniquely suited for success in this context, to broaden the scope of RIC alloBMT with PTCy as a curative therapy for patients with PID/IDS and IBMFS.

This is a Phase II single arm trial to prospectively study a RIC BMT with PTCy to enhance durable engraftment of donor cells and improve outcomes for patients with PID/IDS and IBMFS.

Treatment Plan:

Indwelling central venous catheter Placement of a double lumen central venous catheter will be required for administration of IV medications and transfusion of blood products.

Pre-treatment Evaluation All patients will require documentation of a detailed history and physical examination and standard evaluation of cardiac, pulmonary, liver and renal function. All patients will undergo disease evaluation. Pre-BMT blood will be drawn for correlative labs.

Preparative regimen Alemtuzumab: administered as an IV infusion on days -14 to -12. For patients >10 kg, 3 mg IV test dose over 2 hours followed by 10 mg IV over 2 hours on day -14, 15 mg IV over 2 hours on day -13, and 20 mg IV over 2 hours on day -12. For patients <10 kg, doses are 3 mg, 10 mg, 10 mg, and 10 mg.

Fludarabine: administered as an IV infusion over 30 minutes on days -7 to -3. The dose will be 30 mg/m2/dose (adjusted for renal function).

Melphalan: Recommended to be administered as an IV infusion over 30-60 minutes, depending on volume, on days -3 and -2. The dose will be 70 mg/m2/dose. Alternatively, may be given as 140 mg/m2/dose as a single dose IV infusion per institutional standards on day -2. Other institutional infusion standards are acceptable and will not be a protocol deviation.

Total body irradiation: 200 centigray (cGy) anterior-posterior-posterio-anterior (AP/PA) with 4 megavolt (MV) or 6 MV photons at 8 12 cGy/min at the point of prescription (average separation of measurements at mediastinum, abdomen, and hips) will be administered in a single fraction on day -1. This is only for patients with PID/IDS.

Bone marrow transplantation Bone Marrow will be harvested and infused on day 0. Institutional guidelines for the infusion of bone marrow (i.e. major or minor blood type group (ABO) incompatible bone marrow, etc.) will be followed. The marrow infusion will be done by designated members of the BMT team. The bone marrow graft will not be manipulated to deplete T cells. The donor will be harvested with a target yield of 4 x 10^8 nucleated cells/kg recipient ideal body weight (IBW). The lowest acceptable yield is 2 x 10^8 nucleated cells/kg. The cluster of differentiation (CD)-34+, CD4+, CD8+, and CD3+ cell count in the marrow will be quantified by flow cytometry. Bone marrow graft should be hung to gravity (not infused with a pump). If possible, the total infusion time should be no more than four hours.

GVHD prophylaxis

Post-transplantation Cyclophosphamide (PTCy) Cyclophosphamide (Cy) 50mg/kg will be given on D+3 post-transplant (within 60-72 hr of marrow infusion) and on D+4 post-transplant. Cyclophosphamide will be given as an IV infusion over 1- 2 hours (depending on volume). Dosing of cyclophosphamide is based on ideal body weight for subjects whose ideal body weights less than or equal to subjects' actual body weight. On occasion, a subject's actual body weight may be less than his/her ideal body weight, in which case cyclophosphamide will be dosed using the subject's actual body weight.

Patients will be instructed to increase fluids overnight before cyclophosphamide administration. Hydration with normal saline at 3 cc/kg/hr iv will be started 8 hr prior to cyclophosphamide, then the rate will be reduced to 2 cc/kg/hr for 1 hr pre-cyclophosphamide and continued for at least 8 hr post-cyclophosphamide or administered per institutional standards. Mesna will be given IV at 10 mg/kg/dose concurrent with cyclophosphamide infusion, followed by 40 mg/kg/dose IV over 24 hours, or administered per institutional standards. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of mesna is equal to 100% of the total daily dose of cyclophosphamide.

It is crucial that no immunosuppressive agents are given until 24 hours after the completion of the post-transplant Cyclophosphamide. This includes steroids as anti-emetics. Steroids for disease treatment will attempt to be weaned but are allowed if wean is not possible. Physiologic and stress dose steroids are allowed if necessary. Steroids are allowed as pre-medications if needed.

Tacrolimus On day +5, patients will begin prophylaxis with Tacrolimus (oral (PO) or intravenous (IV) as per institutional standards for starting this prophylaxis).Tacrolimus begins on Day 5, at least 24 hours after completion of post-transplantation Cy. The tacrolimus starting dose will be given per institutional standards for adult or pediatric patients. The recommended, but not required, The starting dose of tacrolimus is 0.015mg/kg IBW/dose IV over 4 hours every 12 hours. , or per institutional standard. Serum trough levels of tacrolimus should be measured around D+7 and the dose should be adjusted based on this level to maintain a level of 5-15 ng/ml. Tacrolimus should be converted to oral dosing when patient has a stable, therapeutic level and is able to tolerate food or other oral medications. For pediatric patients, the oral dosing is approximately two to four times the IV dosing. It is recommended that serum trough levels should be checked at steady state after any dose modification and when switching from IV to oral to ensure therapeutic trough concentrations. Serum trough concentrations should be checked at a minimum weekly thereafter and the dose adjusted accordingly to maintain a level of 5-15 ng/ml. Tacrolimus will be discontinued after the last dose on Day 60 for matched related donors, Day 120 for matched unrelated donors, and day 180 for haploidentical related or mismatched unrelated donors; or may be continued if active GVHD is present. This should be discussed with the PI.

Mycophenolic acid mofetil (MMF) MMF will be given at a dose of 15 mg/kg PO three times daily (TID) (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1 g PO TID). MMF prophylaxis will be discontinued after the last dose on day 35.

Growth factor support Patients will receive Granulocyte-colony stimulating factor (GCSF) (Filgrastim®) 5µg/kg/d subcutaneous (SC) or IV starting at Day 5 and continuing until the absolute neutrophil count (ANC) >1000/mm3 x 3 days. For use in the case of fungal infections or subsequent neutropenia (ANC <500/mm3), GCSF should be continued at the discretion of the treating physician.

Transfusion support Platelet and packed red cell transfusions will be given per current institutional recommendations.

Infection prophylaxis and therapy All infection prophylaxis and therapy will be administered and discontinued as per institutional requirements. The following are recommendations only.

i) During pre-transplant evaluation patients will be screened for respiratory syncytial virus (RSV) and influenza A and B, as well as parainfluenza and other respiratory viruses if symptomatic. Assays of these viruses must be negative for patients to be admitted for transplant. Consideration should be given to institution of antiviral therapy if positive prior to transplant.

ii) Oral hygiene will be maintained according to institutional standards. iii) Antifungal prophylaxis will be administered according to institutional practices. It is important to follow levels of tacrolimus for patients receiving one of the azole antifungal medications. The combination of both drugs can raise the levels of the immunosuppressant to toxic levels. If a patient on tacrolimus is started on an azole antifungal medication, a dose reduction of the tacrolimus is required and levels should be obtained to ensure patients are not in the toxic range.

iv) Pneumocystis jiroveci pneumonia (PJP) prophylaxis will be administered according to institutional practices. Recommendations include administering during the preparative regimen, and then restarting approximately one month post-BMT (or later if white blood cell count (WBC) not recovering) and continuation until at least one year post-BMT.

v) Viral prophylaxis for herpes simplex virus (HSV) and varicella zoster virus (VZV) will be administered according to institutional practices. Recommendations include continuation for at least one year post-BMT and/or while on immunosuppressive medications.

vi) Prophylactic and empiric antibiotics as well as intravenous immunoglobulin (IVIg) will be administered according to institutional practices.

vii) Re-immunization may be performed according to institutional practices.

Anti-ovulatory treatment Menstruating females will are recommended to should be be started on an anti-ovulatory agent, such as Lupron prior to the initiation of the preparative regimen. The treatment administered will be at the discretion of the treating physician.

Post-BMT evaluation Patients will be followed during (i) the initial post-BMT period (ii) after discharge to the referring physician as per standard practice.

ELIGIBILITY:
Inclusion Criteria

Cohort A:

Primary Immune Deficiencies with indication for HCT:

* Chronic granulomatous disease (CGD)
* Wiskott-Aldrich syndrome (WAS)
* Hyper-IgM syndrome
* Common variable immunodeficiency (CVID)
* Leukocyte adhesion deficiency-1 (LAD-1)
* Severe Combined Immunodeficiency (SCID)
* CTLA-4 deficiency
* CARD9 deficiency
* DOCK8 deficiency

Immune Dysregulatory Syndromes:

* Immunodysregulation polyendocrinopathy enteropathy X-linked (IPEX) syndrome
* Hemophagocytic lymphohistiocytosis (HLH) or related disorder with indication for transplant
* CAEBV: Patients with chronic EBV infection (CAEBV) with indication for BMT:

Inherited Bone marrow failure disorders

* Congenital amegakaryocytic thrombocytopenia (CAMT)
* Diamond Blackfan anemia (DBA)
* Shwachman Diamond Syndrome (SDS)
* Thrombocytopenia Absent Radii (TAR)
* Glanzmans thrombasthenia (GT)
* Kostmann syndrome
* Other indications and/or other PID, IDS, and IBMFS diagnoses as deemed appropriate by the PI.

Cohort B: Short telomere syndrome

Cohort C: Confirmed diagnosis of Fanconi anemia or non-Fanconi DNA-dsb repair disorders

* Fanconi anemia
* Non-Fanconi DNA-dsb repair disorders
* Cerunnos-XRCC4-like factor deficiency (XLF or NHEJ1)
* DNA ligase IV deficiency (LIG4)
* Nijmegen breakage syndrome (NBS)
* Increased DNA breakage after exposure of patient cells to DNA cross-linking agents such as diepoxybutane or mitomycin C and germline mutation(s) in an identified Fanconi pathway gene.

Available donor as follows:

* Fully HLA matched sibling or other first-degree family member.
* Fully HLA matched unrelated 10/10 donor using high-resolution DNA-based typing at the following genetic loci: HLA-A, -B, -C, DRB1, and DQB1.
* Mismatched unrelated donor at 8 or 9/10 alleles, using high-resolution typing as above.
* HLA-haploidentical family members of any degree who match at least one allele of each of the following genetic loci: HLA-A, -B, -C, DRB1, and DQB1. A minimum match of 5/10 is therefore required, and will be considered sufficient evidence that the donor and recipient share one HLA haplotype.
* The patient and/or legal guardian must sign informed consent for BMT.
* Patients with adequate organ function as measured by
* Cardiac: Left ventricular ejection fraction (LVEF) at rest must be ≥ 35%. For patients aged <13 years, shortening fraction (SF) > 25% by echocardiogram or LVEF by MUGA may be used.
* Hepatic: Bilirubin ≤ 3.0 mg/dL; and ALT, AST, and Alkaline Phosphatase < 5 x ULN.
* Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or GFR) > 40 mL/min/1.73m2.
* Pulmonary: PFT with FEV1 and FVC >/= 50% of normal and DLCO corrected for Hgb >/= 40% of normal. Patients unable to undergo PFTs should have stable resp status with SaO2 >90% on a max of 2L/min supplemental O2.
* Karnofsky or Lansky performance status ≥70%
* Females and males of childbearing potential must agree to practice 2 effective methods of contraception at the same time, or agree to abstinence.

Exclusion criteria

* Patients will not be excluded on the basis of sex, racial or ethnic background.
* Positive leukocytotoxic crossmatch.
* Prior allogeneic stem cell transplant.
* Uncontrolled bacterial, viral, or fungal infection at the time of enrollment. Uncontrolled is defined as currently taking medication and with progression or no clinical improvement on adequate medical treatment. The investigators recognize that patients with CAEBV may have ongoing EBV viremia at the time of initiating pre-transplant therapy, but other patients should have no uncontrolled bacterial, viral, or fungal infections.
* Diagnosis of idiopathic aplastic anemia
* Seropositivity for the human immunodeficiency virus (HIV)
* Active Hepatitis B or C determined by serology and/or NAT
* Female patients who are diagnosed as pregnant by beta bHCG testing (per institutional practice) or who are breast-feeding.
* Active malignancy or within the timeframe for significant concern for relapse of prior malignancy
* For Cohort B and C: liver biopsy (if performed, not required) with moderate-severe fibrosis/cirrhosis

Donor Eligibility

* Donor must be medically, socially, and psychologically fit to donate
* Bone marrow is the preferred graft source, however, PBSCs may be requested. In particular, PBSCs may be preferred for patients with active viral reactivations and/or for patients who would benefit from a higher count in the graft. Cord blood is not permitted.
* First-degree relatives should be tested for degree of HLA match, CMV serology, ABO type, and complete blood count (CBC). An unrelated donor search should be initiated at the time the patient is referred for BMT.
* Age ≥5 years
* Donors must meet the selection criteria as defined by the Foundation for the Accreditation of Hematopoietic Cell Therapy (FACT).
* Lack of recipient anti-donor HLA antibody in recipient
* Note: In some instances, low level, non-cytotoxic HLA specific antibodies may be permissible if found to be at a level well below that detectable by flow cytometry. This will be decided on a case-by-case basis by the PI and one of the immunogenetics directors.
* In inherited disorders, family members must be tested for carrier and disease status of the underlying disorders. In the event that family members are unaffected carriers, eligibility as donors will be decided upon by the PI on a case-by-case basis
* In the event that two or more eligible donors are identified, the donor will be selected per institutional standards. Suggested criteria include the following:
* Related is preferred over unrelated.
* The potential donor that is youngest in age is preferred.
* For CMV seronegative patients, a CMV seronegative donor is preferred. For CMV seropositive patients, a CMV seropositive donor is preferred.
* Red blood cell compatibility, in order of preference:
* RBC cross match compatible Minor ABO incompatibility, Major ABO incompatibility
* If the patient is male, male donors are preferred.

Ages: 4 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Donor Engraftment | 60 Days
  Rate of donor engraftment ≥95% at day 60 as measured by donor chimerism in whole blood.

SECONDARY OUTCOMES:
Number of patients that have survived at 1 year | 1 year
  Overall Survival (Defined as alive) in patients receiving using reduced intensity conditioning (RIC) hematopoietic stem cell transplant (HSCT) and post-transplant cyclophosphamide (PTCy) for patients with primary immune deficiencies (PID), immune dysregulatory syndromes (IDS), inherited bone marrow failure syndromes (IBMFS), short telomere, Fanconi Anemia and non-Fanconi DNA dsb repair.
Disease Free Survival at 1 year | 1 year
  Disease-Free Survival (defined as without recurrence of underlying disease, without graft failure, and alive) in patients receiving using reduced intensity conditioning (RIC) hematopoietic stem cell transplant (HSCT) and post-transplant cyclophosphamide (PTCy) for patients with primary immune deficiencies (PID), immune dysregulatory syndromes (IDS), inherited bone marrow failure syndromes (IBMFS), short telomere, Fanconi Anemia and non-Fanconi DNA dsb repair.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Symons, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein OR, Bapty S, Lederman HM, Younger MEM, Zambidis ET, Jones RJ, Cooke KR, Symons HJ. Reduced Intensity Bone Marrow Transplantation with Post-Transplant Cyclophosphamide for Pediatric Inherited Immune Deficiencies and Bone Marrow Failure Syndromes. J Clin Immunol. 2021 Feb;41(2):414-426. doi: 10.1007/s10875-020-00898-0. Epub 2020 Nov 6. PMID 33159275